CLINICAL TRIAL: NCT00521898
Title: Prospective Clinical Study on Descemet Membrane Endothelial Keratoplasty (DMEK)
Brief Title: Descemet Membrane Endothelial Keratoplasty (DMEK)
Acronym: DMEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Netherlands Institute for Innovative Ocular Surgery (Other)
Collaborators: Amnitrans Eyebank Rotterdam (Other)
Responsible Party: Principal Investigator, GRJ Melles, MD, PhD, Institute Director, Netherlands Institute for Innovative Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIIOS.2005.14
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Corneal Dystrophies, Hereditary
Keywords: Corneal transplantation, Descemet membrane
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DMEK (Experimental): DMEK as intervention
  Interventions: Procedure: Descemet Membrane Endothelial Keratoplasty (DMEK)

INTERVENTIONS:
Procedure: Descemet Membrane Endothelial Keratoplasty (DMEK)

SUMMARY:
To evaluate isolated Descemet membrane transplantation as a refinement of previous advanced techniques for corneal transplantation, like Descemet Stripping Endothelial Keratoplasty (DSEK)

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Corneal endothelial disorders

Exclusion Criteria:

* N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2005-02; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Best spectacle corrected visual acuity | 2005-2015

SECONDARY OUTCOMES:
Corneal endothelial cell density | 2005-2015

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit R Melles, MD, PhD, Principal Investigator — Netherlands Institute for Innovative Ocular Surgery
Locations (1):
- Netherlands Institute for Innovative Ocular Surgery, Rotterdam, Netherlands

REFERENCES:
- [Background] Birbal RS, Baydoun L, Ham L, Miron A, van Dijk K, Dapena I, Jager MJ, Bohringer S, Oellerich S, Melles GRJ. Effect of Surgical Indication and Preoperative Lens Status on Descemet Membrane Endothelial Keratoplasty Outcomes. Am J Ophthalmol. 2020 Apr;212:79-87. doi: 10.1016/j.ajo.2019.12.011. Epub 2019 Dec 18. PMID 31863726
- [Background] Birbal RS, Ni Dhubhghaill S, Bourgonje VJA, Hanko J, Ham L, Jager MJ, Bohringer S, Oellerich S, Melles GRJ. Five-Year Graft Survival and Clinical Outcomes of 500 Consecutive Cases After Descemet Membrane Endothelial Keratoplasty. Cornea. 2020 Mar;39(3):290-297. doi: 10.1097/ICO.0000000000002120. PMID 31478948
- [Background] Rodriguez-Calvo-de-Mora M, Quilendrino R, Ham L, Liarakos VS, van Dijk K, Baydoun L, Dapena I, Oellerich S, Melles GR. Clinical outcome of 500 consecutive cases undergoing Descemet's membrane endothelial keratoplasty. Ophthalmology. 2015 Mar;122(3):464-70. doi: 10.1016/j.ophtha.2014.09.004. Epub 2014 Oct 22. PMID 25439596
- [Background] Vasiliauskaite I, Oellerich S, Ham L, Dapena I, Baydoun L, van Dijk K, Melles GRJ. Descemet Membrane Endothelial Keratoplasty: Ten-Year Graft Survival and Clinical Outcomes. Am J Ophthalmol. 2020 Sep;217:114-120. doi: 10.1016/j.ajo.2020.04.005. Epub 2020 Apr 10. PMID 32283096
- [Result] Melles GR, Ong TS, Ververs B, van der Wees J. Descemet membrane endothelial keratoplasty (DMEK). Cornea. 2006 Sep;25(8):987-90. doi: 10.1097/01.ico.0000248385.16896.34. PMID 17102683
- [Result] Melles GR. Posterior lamellar keratoplasty: DLEK to DSEK to DMEK. Cornea. 2006 Sep;25(8):879-81. doi: 10.1097/01.ico.0000243962.60392.4f. No abstract available. PMID 17102659
- [Derived] Dirisamer M, Yeh RY, van Dijk K, Ham L, Dapena I, Melles GR. Recipient endothelium may relate to corneal clearance in descemet membrane endothelial transfer. Am J Ophthalmol. 2012 Aug;154(2):290-296.e1. doi: 10.1016/j.ajo.2012.02.032. Epub 2012 May 23. PMID 22633346
- [Derived] Naveiras M, Dirisamer M, Parker J, Ham L, van Dijk K, Dapena I, Melles GR. Causes of glaucoma after descemet membrane endothelial keratoplasty. Am J Ophthalmol. 2012 May;153(5):958-966.e1. doi: 10.1016/j.ajo.2011.10.003. Epub 2012 Jan 28. PMID 22285014
- [Derived] Dirisamer M, van Dijk K, Dapena I, Ham L, Oganes O, Frank LE, Melles GR. Prevention and management of graft detachment in descemet membrane endothelial keratoplasty. Arch Ophthalmol. 2012 Mar;130(3):280-91. doi: 10.1001/archophthalmol.2011.343. Epub 2011 Nov 14. PMID 22084160
- [Derived] Dirisamer M, Ham L, Dapena I, Moutsouris K, Droutsas K, van Dijk K, Frank LE, Oellerich S, Melles GR. Efficacy of descemet membrane endothelial keratoplasty: clinical outcome of 200 consecutive cases after a learning curve of 25 cases. Arch Ophthalmol. 2011 Nov;129(11):1435-43. doi: 10.1001/archophthalmol.2011.195. Epub 2011 Jul 11. PMID 21746971
- [Derived] Dirisamer M, Dapena I, Ham L, van Dijk K, Oganes O, Frank LE, van der Wees J, Melles GR. Patterns of corneal endothelialization and corneal clearance after descemet membrane endothelial keratoplasty for fuchs endothelial dystrophy. Am J Ophthalmol. 2011 Oct;152(4):543-555.e1. doi: 10.1016/j.ajo.2011.03.031. Epub 2011 Jul 2. PMID 21726849
- [Derived] Dapena I, Ham L, Moutsouris K, Melles GR. Incidence of recipient Descemet membrane remnants at the donor-to-stromal interface after descemetorhexis in endothelial keratoplasty. Br J Ophthalmol. 2010 Dec;94(12):1689-90. doi: 10.1136/bjo.2010.186189. Epub 2010 Aug 1. No abstract available. PMID 20679083
- [Derived] Dapena I, Ham L, van Luijk C, van der Wees J, Melles GR. Back-up procedure for graft failure in Descemet membrane endothelial keratoplasty (DMEK). Br J Ophthalmol. 2010 Feb;94(2):241-4. doi: 10.1136/bjo.2009.160945. Epub 2009 Aug 26. PMID 19713195
- [Derived] Ham L, van Luijk C, Dapena I, Wong TH, Birbal R, van der Wees J, Melles GR. Endothelial cell density after descemet membrane endothelial keratoplasty: 1- to 2-year follow-up. Am J Ophthalmol. 2009 Oct;148(4):521-7. doi: 10.1016/j.ajo.2009.04.025. Epub 2009 Jun 25. PMID 19555921
- [Derived] Balachandran C, Ham L, Verschoor CA, Ong TS, van der Wees J, Melles GR. Spontaneous corneal clearance despite graft detachment in descemet membrane endothelial keratoplasty. Am J Ophthalmol. 2009 Aug;148(2):227-234.e1. doi: 10.1016/j.ajo.2009.02.033. Epub 2009 May 13. PMID 19442962
- [Derived] Ham L, Balachandran C, Verschoor CA, van der Wees J, Melles GR. Visual rehabilitation rate after isolated descemet membrane transplantation: descemet membrane endothelial keratoplasty. Arch Ophthalmol. 2009 Mar;127(3):252-5. doi: 10.1001/archophthalmol.2008.619. PMID 19273786